CLINICAL TRIAL: NCT02516891
Title: Jailed Wire Technique in the Treatment of Coronary Bifurcations Lesions With Stent: Prospective Randomized Study With Stereoscopic Microscopy
Brief Title: Jailed Wire Technique in the Treatment of Coronary Bifurcations Lesions With Stent: Stereoscopic Microscopy Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PI12/00440
Record Dates: First submitted 2014-07-23; First posted 2015-08-06 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Coronary Health Disease
Keywords: treatment; stent; coronary bifurcations lesions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- hydrophilic wire/Drug-Eluting Stents (Experimental): Will include 100 patients with coronary bifurcation lesions in that they will be treated with stents and in which the technique is used jailed guide.
  Interventions: Device: Drug-Eluting Stents implantation in bifurcation lesions
- Non hydrophilic wire/Drug-Eluting Stents (No Intervention): Will include 100 patients with coronary bifurcation lesions in that they will be treated with stents and in which the technique is used jailed guide.non hydrophilic guide.

INTERVENTIONS:
Device: Drug-Eluting Stents implantation in bifurcation lesions
  Arms: hydrophilic wire/Drug-Eluting Stents

SUMMARY:
The aims of this study are: 1) To identify more resistant the guidewire type to the retrieval maneuvers after the jailing.

2) To determined anatomic and technical factors influencing the induced damage in the guidewire.

Design of the study: prospective randomized study to compare 2 types of guidewire: hydrophilic and no hydrophilic. Patients and methods: Two hundred patients with bifurcation coronary lesions will be included. All of then will be treated by provisional side-branch stenting using the jailed wire technique. One hundred patients will be randomized to hydrophilic wires and another 100 patients to non-hydrophilic wires.

DETAILED DESCRIPTION:
The percutaneous approach of bifurcation lesions is a complex procedure; when the stent is implanted at main vessel, a closure of the side-branch may occur. The re-wiring of the side-branch in these conditions may be difficult or even impossible. To facilitate the re-wiring maneuvers the operators use the jailed wired technique. For this technique a guide-wire is introduced in the side-branch before main vessel stent implantation; after the stent deployment the wire remains jailed between the vessel wall and the metallic structure of the stent. If the side-branch became occluded, this wire is a good landmark of it is position, facilitating the access with a new wire. However, the rupture of the wire has been described in some cases, during the retrieval maneuvers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with atherosclerotic coronary disease and bifurcation lesions requiring protection with side branch.
* The art of imprisoned guide.
* The main branch should be greater than 2.5 mm in diameter at the operator's visual estimate.
* The side branch must exceed 2 mm in diameter or have sufficient authority to protect the operator decides with a guide for the release of the main vessel stent.
* Patients with the above characteristics and main or side branch of any length.
* Patients with bifurcation lesions with any morphology of the Medina classification: 1 1 1 1 0 1 0 1 1, 110, 001, 010, 100.
* Treatment of bifurcation with any technique and any type of stent in the side branch meets the criteria above.
* Symptoms of stable angina or acute coronary syndrome.

Exclusion Criteria:

* Patients with collateral bouquet of little significance.
* Patients in cardiogenic shock.
* Patients in whom it is impossible to guide the placement of the side branch before implantation in the glass principal.
* Patients who do not give their consent for the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2012-02; Primary Completion 2015-06 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
No damage: the guidewire suffered no loss of integrity over its entire length | 3 years
Slight damage: the external cover suffered loss of integrity < 2 mm | 3 years
Moderate damage: the external cover suffered loss of integrity > 2 mm | 3 years
Severe damage: visible changes to the inner cover of the guidewire. | 3 years
Fracture: discontinuity at some point along the guidewire | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Reina Sofía, Córdoba, Córdoba, Spain

REFERENCES:
- [Derived] Pan M, Ojeda S, Villanueva E, Chavarria J, Romero M, Suarez de Lezo J, Mazuelos F, Segura J, Carrasco F, Hidalgo F, Lopez Aguilera J, Rodriguez S, Puente M, Suarez de Lezo J. Structural Damage of Jailed Guidewire During the Treatment of Coronary Bifurcation Lesions: A Microscopic Randomized Trial. JACC Cardiovasc Interv. 2016 Sep 26;9(18):1917-24. doi: 10.1016/j.jcin.2016.06.030. PMID 27659568